CLINICAL TRIAL: NCT00340301
Title: Exposure to Neurotoxins as Risk Factors for ALS: Measurement of Genes, Proteins, Neurotoxicants, and Other Factors Potentially Associated With ALS
Brief Title: Exposure to Neurotoxins as Risk Factors for ALS
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999903210; 03-E-N210
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2019-01-25 (Actual); Status verified 2019-01-23

CONDITIONS: ALS
Keywords: Polymorphism; Neurodegenerative Diseases; ALS
MeSH Terms: conditions — Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

SUMMARY:
Chemicals called neurotoxins can harm the nervous system. Amyotrophic lateral sclerosis (ALS) is a progressive disease affecting movement. Researchers have studied many possible causes of ALS, including injury, diet, and exposure to chemicals, but these studies were inconclusive.

The purpose of this study was to determine whether exposure to lead or other neurotoxins can contribute to ALS. The study also evaluated lifestyle and dietary patterns. The study was completed in 1994-1996.

One hundred eighty-two participants took part in this study 110 patients with ALS and 72 who did not have ALS. Each completed a questionnaire concerning lifestyle, diet, and residential, job, and medical history. Participants contributed 50 cc of blood, used to measure lead, as well as clippings of their toenails, used to measure mercury and other metals. They then underwent an XRF test (an X-ray procedure) to measure the level of lead in their shinbones and knees. Genes related to ALS or susceptibility to lead exposure were also evaluated.

DETAILED DESCRIPTION:
OBJECTIVES: Stored blood and toenail samples are available from a case-control study of ALS conducted in 1993-1996. The purpose of the initial study was to examine the relationship to ALS of lead and other exposures, including mercury, pesticides, and solvents, as well as genetic susceptibility to these exposures. The protocol was closed in May 1997 (closed protocol #95-007) after recruitment of study subjects ended. The objective of the present proposal is to reopen the protocol to permit measurement in blood or toenails of genes, proteins, neurotoxicants, and other factors or agents potentially associated with ALS, as well as analyses of existing data. The short-term goal is to measure (i) polymorphisms in DNA repair genes; (ii) serum protein profiles; and (iii) serum organochlorine pesticide levels. Other factors may be of interest in the future, for example polymorphisms in other genes or levels of metals in blood or toenails. We also plan (iv) to continue analyses of existing data. Some data analysis will involve combining data from the original ALS study with data from the Harvard Normative Aging Study, a cohort study of World War II verterans that has collected demographic, lifestyle, and medical data as well as information on bone and blood lead levels.

STUDY POPULATION: No new subjects will be recruited for this protocol. The original study involved 110 ALS cases, 31 hospital controls with other neurologic diseases, and 256 population controls, recruited in New England between 1993 and 1996. The population controls were frequency matched to the cases on the basis of age, gender, race, and region within New England.

DESIGN: The original study was a case-control study. Data collection involved an interview collection of blood and toenail samples, and measurement of bone lead using x-ray fluorescence. Stored blood and/or toenail samples are available from 107 ALS cases, 31 hospital controls, and 39 population controls. The present study will use conventional techniques to measure genetic polymorphisms and serum organochlorine levels and newly developed SLDI-TOF technology to evaluate serum protein profiles.

OUTCOME PARAMETERS: The outcome parameter is risk of ALS. Associations with ALS risk will be evaluated for polymorphisms in DNA repair genes; serum protein profiles; and organochlorine pesticide levels in serum.

ELIGIBILITY:
* INCLUSION CRITERIA:

Cases were eligible to participate in the original study if (1) they had received a diagnosis of ALS within 2 years; (2) they lived in New England at least half the year; (3) they spoke English; (4) they were mentally and physically able to participate. The same inclusion criteria were used for controls.

EXCLUSION CRITERIA:

Potential controls were excluded if they had a physician diagnosis of a neurodegenerative disease, polio, post-polio syndrome, or nondiabetic neuropathy.

Pregnant women were excluded from both case and control groups.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2003-06-03; Study Completion 2019-01-23

PRIMARY OUTCOMES:
Measurement in blood or toenails of genes, proteins, neurotoxicants, and other factors or agents potentially associated with ALS

CONTACTS AND LOCATIONS:
Overall Officials: Freya Kamel, Ph.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- New England Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Nelson LM. Epidemiology of ALS. Clin Neurosci. 1995-1996;3(6):327-31. PMID 9021253
- [Background] Shaw PJ. Motor neurone disease. BMJ. 1999 Apr 24;318(7191):1118-21. doi: 10.1136/bmj.318.7191.1118. No abstract available. PMID 10213726
- [Background] Mitchell JD. Amyotrophic lateral sclerosis: toxins and environment. Amyotroph Lateral Scler Other Motor Neuron Disord. 2000 Sep;1(4):235-50. doi: 10.1080/14660820050515061. PMID 11465017